CLINICAL TRIAL: NCT01530711
Title: Treatment of Hepatorenal Syndrome With Terlipressin Infusion Adjusted to Hemodynamic Response
Acronym: AMELIORATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pere Gines (Other)
Responsible Party: Sponsor-Investigator, Pere Gines, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMELIORATE
Record Dates: First submitted 2012-02-09; First posted 2012-02-10 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Cirrhosis; Hepatorenal Syndrome Type I
MeSH Terms: conditions — Fibrosis | interventions — Terlipressin; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- terlipressin (Experimental)
  Interventions: Drug: Terlipressin and albumin

INTERVENTIONS:
Drug: Terlipressin and albumin — Terlipressin dose: 2mg/24h, it will be modified depending on: Arterial pressure increase < 10 mmHg and the creatinine values decrease <25%, it will be increased every 8 hours until reaching an increase of at least 10mmHg arterial pressure or a creatinine decrease of the 25%.
  Albumin: Initial dose (first day) of 1g/Kg (up to a maximum of 100g) and the following days from 20 to 40 g/day.

SUMMARY:
Observe the effect of terlipressin on renal function in patients with SHR type I adjusting the dose based on hemodynamic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatorenal syndrome type 1.
* Signed informed consent.
* No exclusion criteria.
* At least 18 years old
* Negative pregnancy test in serum or urine in women of childbearing age, and agree to use adequate contraception since at least 14 days prior to the first dose of study drug until 14 days after the last.

Exclusion Criteria:

* Hepatocellular carcinoma: exclusion of patients with hepatocellular carcinoma who present more than 3 nodules, single nodule larger than 5 cm, tumor portal thrombosis or extrahepatic tumor spread.
* Active bacterial infection with symptoms of systemic inflammatory response (fever, tachycardia, tachypnea, hypotension, septic or blood count).
* Cardiac or respiratory failure clinically significant.
* Clinically significant peripheral artery disease.
* A history of ischemic heart disease.
* Hypersensitivity to terlipressin and / or albumin or any of the excipients.
* Pregnancy.
* Septic shock.
* Chronic renal failure.
* Women in lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in arterial pressure and creatinine | 4 months

SECONDARY OUTCOMES:
Changes in plasmatic renin activity and aldosterone and noradrenaline concentration. | 4 months
Treatment-related adverse events | 4 months
Hepatorenal Syndrome reversion due to hemodynamic changes. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: German Soriano Pastor, MD, Principal Investigator — gsoriano@santpau.cat; Juan Cordoba, MD, Principal Investigator — jcordoba@vhebron.net; Isabel Cirera Lorenzo, MD, Principal Investigator — ICirera@parcdesalutmar.cat; Marta Martín Llahí, MD, Principal Investigator — martinllahi@gmail.com; Jordi Sánchez Delgado, MD, Principal Investigator — jsanchezd@tauli.cat
Locations (6):
- Spain (6):
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall d´Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Moisés Broggi, Sant Joan Despí, Barcelona